CLINICAL TRIAL: NCT01511835
Title: Efficacy of Myo-inositol in Preventing Gestational Diabetes in High-risk Pregnant Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: MyoIN_diab
Record Dates: First submitted 2011-11-16; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Gestational Diabetes
Keywords: diabetes; pregnancy; myo-inositol
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Inositol; Folic Acid

ARMS (3):
- Myo-inositol powder (Experimental)
  Interventions: Dietary Supplement: inositol + folic acid
- Myo-inositol soft gel capsules (Experimental)
  Interventions: Dietary Supplement: inositol + folic acid
- Folic acid (Placebo Comparator)
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Dietary Supplement: inositol + folic acid — 2000 mg of inositol+200mcg of folic acid; 2 per diem
  Arms: Myo-inositol powder
Dietary Supplement: inositol + folic acid — 600 mg of inositol + 200mcg of folic acid; 2 cp per diem
  Arms: Myo-inositol soft gel capsules
Drug: Folic Acid — Folic Acid 400mcg; 1 cp/die
  Arms: Folic acid

SUMMARY:
The aim of this study is to evaluate the efficacy of myo-inositol in preventing gestational diabetes in high risk pregnant women.

ELIGIBILITY:
Inclusion Criteria:

60 women in their first trimester of pregnancy affected by one or more of the following risk factors:

* Glycemia levels > 92 mg/dl
* BMI > 30
* At least a parent or a brother (or sister)affected by diabetes
* Pre-existing pregnancy with gestational diabetes

Exclusion Criteria:

* Pregnant women affected by pregestational diabetes
* Twin pregnancy
* Patients affected by pre-existing diseases in pregnancy (diabetes excluded)
* Patients affected by chronic disorders

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult

PRIMARY OUTCOMES:
OGTT
  The diagnostic 75g oral glucose tolerance test (OGTT) is performed between 24 and 28 weeks of gestation.

SECONDARY OUTCOMES:
Number of pregnant women with gestational diabetes
Number of pregnant women requiring insulin treatment
Weight gain at the end of pregnancy
Number of newborn infants whose weight is more than 4000 g
Number of newborn infants requiring Neonatal Intensive Care (NIC)

CONTACTS AND LOCATIONS:
Locations (1):
- AGUNCO, Rome, Italy

REFERENCES:
- [Background] Papaleo E, Unfer V, Baillargeon JP, Chiu TT. Contribution of myo-inositol to reproduction. Eur J Obstet Gynecol Reprod Biol. 2009 Dec;147(2):120-3. doi: 10.1016/j.ejogrb.2009.09.008. Epub 2009 Oct 2. PMID 19800728
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Derived] Motuhifonua SK, Lin L, Alsweiler J, Crawford TJ, Crowther CA. Antenatal dietary supplementation with myo-inositol for preventing gestational diabetes. Cochrane Database Syst Rev. 2023 Feb 15;2(2):CD011507. doi: 10.1002/14651858.CD011507.pub3. PMID 36790138